CLINICAL TRIAL: NCT05356507
Title: The Effects of Spiritual Needs on Spiritual Well-Being in Patients With Brain Tumors: A Structural Equation Modeling Approach
Status: Withdrawn | Type: Observational
Why Stopped: 0 accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0878; NCI-2021-12910 (Other: NCI-CTRP Clinical Trials Reporting Process)
Record Dates: First submitted 2022-04-11; First posted 2022-05-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patient population — Questionnaires, standard of care

SUMMARY:
The aim of this study is to describe a patient's Spiritual Needs and related factors that contribute to a patient's Spiritual Well-Being in the context of perioperative care.

The primary objective of this study is to examine the fit of the Structural Equation Model (SEM) of the theory on Spiritual Well-Being (SWB) and explain how SWB is affected by Symptom Burden (SB), Psychological Distress (PsD), and Spiritual Needs (SN) reported by the patients with brain tumors before having surgery.

DETAILED DESCRIPTION:
The aim of this study is to describe a patient's Spiritual Needs and related factors that contribute to a patient's Spiritual Well-Being in the context of perioperative care.

The primary objective of this study is:

To examine the fit of the Structural Equation Model (SEM) of the theory on Spiritual Well-Being (SWB) and explain how SWB is affected by Symptom Burden (SB), Psychological Distress (PsD), and Spiritual Needs (SN) reported by the patients with brain tumors before having surgery.

This study will address the following secondary objectives:

1. To examine bivariate relationships between SB, PsD, and SN.
2. To explore effects of patients' spirituality on the relationship between patients' SN and SWB.

This study is not powered to test hypotheses concerning the secondary objectives but will specifically examine through descriptive statistics and confidence intervals the following:

1. SN, PsD, and SB are positively correlated with each other.
2. SN negatively influences SWB.
3. SN positively influences spirituality.
4. Spirituality positively influences SWB.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients at MDACC who are 18 years or older;
* Are being/have been seen at the MD Anderson Neurosurgery clinic;
* Have a diagnosis of a primary or metastatic intracranial or skull-based brain, pituitary, or meningeal lesions;
* Are scheduled to undergo surgical intervention.

Exclusion Criteria:

* Have preferred language listed other than English on the chart;
* Present with cognitive functional impairment, evidence of expressive or receptive aphasia, or gross dysfunction limiting memory or ability to complete a self-report questionnaire, which will be determined by reviewing provider's notes;
* Refusal to participate in research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a diagnosis of primary or metastatic brain tumors who are scheduled to undergo surgical interventions
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the Spiritual Needs on Spiritual Well-Being in Patients with Brain Tumors, utilizing the Structural Equation Model (SEM) of the theory on Spiritual Well-Being (SWB). | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anecita Fadol, BLS, MSN, PHD, RN, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org